CLINICAL TRIAL: NCT04303325
Title: Effect of Esketamine on Postoperative Depression、Gut Microbiota、Bispectral Index Data of Depression Patients Undergoing Breast Cancer Operation (ESPOD-BI)
Acronym: ESPOD-BI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenfei Tan, Professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200225
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Depression
Keywords: depression; sleep deprivation; gut microbiota; bispectral index
MeSH Terms: conditions — Depression; Sleep Deprivation | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): All depression patients undergoing breast cancer operation will be to the treatment intervention with general anesthesia as an adjunct to saline.
  Interventions: Drug: Saline Solution
- Esketamine (Active Comparator): All depression patients undergoing breast cancer operation will be to the treatment intervention with general anesthesia as an adjunct to esketamine.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Esketamine — All depression patients undergoing breast cancer operation will be to the treatment intervention with general anesthesia as an adjunct to esketamine 0.2mg/kg.
  Arms: Esketamine
Drug: Saline Solution — All depression patients undergoing breast cancer operation will be to the treatment intervention with general anesthesia as an adjunct to saline.
  Arms: Control

SUMMARY:
This study is a prospective, randomized, controlled (randomized, parallel group, concealed allocation), double-blinded trial. All depression patients undergoing breast cancer operation will be randomized 1:1 to the treatment intervention with general anesthesia as an adjunct to esketamine or saline. The objective of the trial is to evaluate the postoperative depression、gut microbiota、bispectral index data of patients undergoing breast cancer operation with esketamine or saline.

DETAILED DESCRIPTION:
For female patients, breast cancer patients have a high risk of developing depression, and approximately 20%-45% of breast cancer patients suffer from postoperative depression. Esketamine is an anesthetic in analgesia, and has presently become more and more popular for treating anti-depression, particularly for resistant depression.

This study is a prospective, randomized, controlled (randomized, parallel group, concealed allocation), double-blinded trial. All depression patients undergoing breast cancer operation will be randomized 1:1 to the treatment intervention with general anesthesia as an adjunct to esketamine or saline. The objective of the trial is to evaluate the postoperative depression、gut microbiota、bispectral index data of patients undergoing breast cancer operation with esketamine or saline

ELIGIBILITY:
Inclusion Criteria:

* At least18 years and pre-menopausal;
* scheduled to undergo elective breast cancer operation;
* American Society of Anaesthesiologists (ASA) risk classification I-II.
* Montgomery-asberg Depression Rating Scale (MADRS) score ≥22

Exclusion Criteria:

* Cognitive difficulties
* Partial or complete gastrectomy
* Previous esophageal surgery
* Inability to conform to the study's requirements
* Ongoing participation or participation in another study <1 month ago

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 72 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-asberg Depression Rating Scale score | from baseline to postoperative 24 hours
  Changes of Montgomery-asberg Depression Rating Scale score

SECONDARY OUTCOMES:
Bispectral index | from 8pm to 6am on the first postoperative night
  Changes of bispectral index data
Gut microbiota | from baseline to postoperative 72 hours
  changs of gut microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No